CLINICAL TRIAL: NCT04341688
Title: A Double Blind, Randomized Controlled Pilot Trial of Gargling Agents in Reducing Intraoral Viral Load Among Laboratory Confirmed COVID-19 Patients: GARGLES STUDY
Brief Title: A Clinical Trial of Gargling Agents in Reducing Intraoral Viral Load Among COVID-19 Patients
Acronym: GARGLES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, BDS, MS, FCPS, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020-Sur-ERC-4926
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Covid-19
Keywords: Covid-19;; coronavirus disease; povidone; hydrogen peroxide; neem extracts; topical therapy; gargle
MeSH Terms: conditions — COVID-19 | interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: A quadruple blind randomized controlled trial followed by laboratory based analysis. Six parallel groups of participants using various gargles and nasal lavage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical colored and shaped bottles containing different study drugs. This will be provided by the pharmacy services of the university hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Povidone-Iodine 0.2% (BETADINE®) (Experimental): 0.2% Povidone-Iodine (BETADINE®) 10 ml gargle and nasal lavage for 20-30 seconds, thrice daily for 6 days.
  Interventions: Drug: Gargle/Mouthwash
- Hydrogen peroxide 1% (ActiveOxy) (Experimental): ActiveOxy (1% Hydrogen peroxide) 10 ml gargle and nasal lavage for 20-30 seconds, thrice daily for 6 days.
  Interventions: Drug: Gargle/Mouthwash
- Neem extract (Azadirachta indicia) (Active Comparator): Neem extract (Azadirachta indicia) gargle will be prepared by chemistry laboratory. patients will do 10ml gargle and nasal lavage for 20-30 seconds, thrice daily for 6 days.
  Interventions: Drug: Gargle/Mouthwash
- Hypertonic saline (2%NaCl) (Active Comparator): 10 ml gargle and nasal lavage using Hypertonic saline for 20-30 seconds, thrice daily for 6 days.
  Interventions: Drug: Gargle/Mouthwash
- Positive controls (Placebo Comparator): 10 ml gargle and nasal lavage using distilled water for 20-30 seconds, thrice daily for 6 days.
  Interventions: Drug: Gargle/Mouthwash

INTERVENTIONS:
Drug: Gargle/Mouthwash — There will be 50 patients in six study groups. Group A (n=10) patients on 10 ml gargle and nasal lavage using 0.2% Povidone-Iodine (Betadiene®) for 20-30 seconds, thrice daily for 6 days.
  Group B (n=10) patients will be subjected to 10 ml gargle and nasal lavage using 1% Hydrogen peroxide (ActiveOxy®) for 20-30 seconds, thrice daily for 6 days.
  Group C will comprised of (n=10) subjects on 10ml gargle and nasal lavage using Neem extract solution (Azardirachta indica) formulated locally) for 20-30 seconds, thrice daily for 6 days.
  Group D (n=10) patients will use 2% hypertonic saline (Plabottle®) gargle and nasal lavage for a similar time period.
  Group E (n=10) will serve as positive controls. These will be given simple distilled water gargles and nasal lavage for 20-30 seconds, thrice daily for six days Whereas Group F (n=5) will comprise of negative controls, who will not use any gargles or nasal lavage during study period.
  Other Names: Gargling agent; Mouthrinse

SUMMARY:
Pakistan is a resource restraint country, it's not possible to carry out coronavirus testing at mass scale. Simple cost effective intervention against the present pandemic is highly desirable.

For patients: Identifying an antiviral gargle that could substantially reduce the colonies of COVID-19 residing in mouth and oro-naso-pharynx is likely to reduce the viral load. Such reduction in the viral load through surface debridement could aid the effective immune response in improving the overall symptoms of the patients.

For dentists: This study is important because the nature of the dental profession involves aerosol production, carrying out dental work on asymptomatic patients carrying coronavirus puts the entire dental team at a great risk of not only acquiring the infection but also transmitting it to the others. Antiviral gargles could be used by dentist and their auxiliaries as prophylaxis.

For physicians and nurses: The risk of morbidity and mortality is high among physicians and nurses involved in the screening and management of Covid-19 patients. Globally, over 215 physicians and surgeons have died while taking care of Covid-19 patients. The cause of death is attributed to high exposure of viral load. The antiviral gargles and nasal lavage can decrease the fatalities among doctors and nurses.

Thus, patients, physicians, nurses and dentists, all could be benefited with this findings of this study.

DETAILED DESCRIPTION:
It will be a parallel group, quadruple blind-randomized controlled pilot trial annexed with a laboratory based study. Clinical trial will be carried out at the Aga Khan University Hospital (AKUH), Karachi, Pakistan. Patients will be inducted from the pool of known patients (laboratory confirmed COVID-19 participants) within 7 days of the onset of viral infection symptoms, already admitted at AKUH. Molecular and immunological testing will be done at the Juma laboratory of AKUH. The intervention drugs (Povidone-Iodine, Hydrogen Peroxide and Hypertonic Saline will be obtained from the AKUH distribution department and/ or AKUH pharmacy. The Neem extract will be compounded at the Chemistry department, University of Karachi/ HEJ institute of Organic Chemistry, University of Karachi.

We will need 50 patients. There will be five study groups. Group A (n=10) patients on 10 ml gargle and nasal lavage with of 0.2% Povidone-Iodine for 20-30 seconds, twice daily for 5 days. Group B (n=10) patients will be subjected to 10 ml gargle and nasal lavage with 1% Hydrogen peroxide for 20-30 seconds, twice daily for 5 days. Group C will comprise of (n=10) subjects using 10ml gargle and nasal lavage with Neem extract (Azardirachta indica) for 20-30 seconds, twice daily for 5 days. Group D (n=10) patients will use 2% hypertonic saline gargle and nasal lavage for a similar time period. Group E (n=10) will serve as positive controls. These will be given simple distilled water gargles and nasal lavage for 20-30 seconds, thrice daily for six days. For nasal lavage, a special douche syringe will be provided to each participant. Its use will be thoroughly explained by the data collection officer.

Data collection: The baseline oral swab will be taken from the posterior pharyngeal wall/ tonsillar area on day one before initiating the gargles by trained dentist. The end-point oral swab will be taken on day 7, just after using the prescribed gargle. Patient will be provided with a special hood so that they themselves don't generate aerosol in the immediate vicinity while carrying out the gargling and nasal lavage.

Data will be analyzed using SPSS for Windows (version 23.0 SPSS) and Graph Pad Prism 7.0 software.

Mean and standard deviation of the continuous variables (age, COVID-19 viral counts and cytokine profiles at baseline and endpoint etc.) will be computed. Frequency distribution of the categorical variables will be determined (gender, co-morbids, presence of hypertension, diabetes, periodontal status etc.) Repeated measures ANOVA will be used to compare the reduction in intra-oral viral load and the changes in the inflammatory biomarkers in the study groups. In case of substantially low count of participants in the study groups, non-parametric tests such as Kruskal-Wallis or Friedman test will be employed. Multiple linear regression (MLR) will done to predict changes in the Covid-19 viral load and cytokine profiles. A subset analysis using Zero inflated negative binomial (ZINB) model will be employed, provided a significant reduction in viral load is observed in any of the study groups. A p-value of <0.05 will be taken as statistically significant. {20a}

The biases and confounders can be taken care at following four levels:

At recruitment stage, we will use restriction i.e. only those COVID positive subjects will be recruited who have no other major co-morbidities. At intervention assignment, the random group allocation will ensure even distribution of the confounders in the study groups thus their differential effect on the outcome will be addressed. At analysis, we will employ regression analysis (as described above) to account for biases and confounders and lastly, the subset analysis will stratify the data and nullify the effect of biases.

Interim analysis {20b} is not planned on account of a short duration of the study. Missing data/ uncompliant patients {20c} will be omitted from the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are laboratory confirmed Covid-19 positive male or female subjects in the age range of 18-65 years, within seven days of the onset of mild to moderate symptoms of viral infection, already admitted in the hospital.

Exclusion Criteria:

* Edentulous patients, patients with low Glasgow coma score, intubated, immune-compromised, history of radiotherapy or chemotherapy will be excluded. Patients with known pre-existing chronic mucosal lesions such as lichen planus will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Intraoral viral load | Five days of using gargles
  Intraoral viral load as deciphered by RT-PCR

SECONDARY OUTCOMES:
Salivary cytokine profile | Five days of using gargles
  Salivary cytokine profiles of IL-2, IL-4, IL-6, IL-10, TNF-α, IFN-γ and IL-17.

CONTACTS AND LOCATIONS:
Overall Officials: Syed MR Kazmi, FCPS, Study Director — Aga Khan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Background] Shafiq HB, Amin U, Nawaz S. Comparative analysis of various antimicrobial agents present in locally available mouthwashes against oral pathogens. Pak J Pharm Sci. 2018 Sep;31(5):1881-1887. PMID 30150184
- [Background] Tanzer JM, Slee AM, Kamay BA. Structural requirements of guanide, biguanide, and bisbiguanide agents for antiplaque activity. Antimicrob Agents Chemother. 1977 Dec;12(6):721-9. doi: 10.1128/AAC.12.6.721. PMID 931371
- [Background] Lai P, Coulson C, Pothier DD, Rutka J. Chlorhexidine ototoxicity in ear surgery, part 1: review of the literature. J Otolaryngol Head Neck Surg. 2011 Dec;40(6):437-40. PMID 22420428
- [Background] Hirata K, Kurokawa A. Chlorhexidine gluconate ingestion resulting in fatal respiratory distress syndrome. Vet Hum Toxicol. 2002 Apr;44(2):89-91. PMID 11931511
- [Background] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Background] Tiwari V, Darmani NA, Yue BY, Shukla D. In vitro antiviral activity of neem (Azardirachta indica L.) bark extract against herpes simplex virus type-1 infection. Phytother Res. 2010 Aug;24(8):1132-40. doi: 10.1002/ptr.3085. PMID 20041417
- [Background] Ahmad A, Javed MR, Rao AQ, Husnain T. Designing and screening of universal drug from neem (Azadirachta indica) and standard drug chemicals against influenza virus nucleoprotein. BMC Complement Altern Med. 2016 Dec 16;16(1):519. doi: 10.1186/s12906-016-1469-2. PMID 27986088
- [Background] Ramalingam S, Graham C, Dove J, Morrice L, Sheikh A. A pilot, open labelled, randomised controlled trial of hypertonic saline nasal irrigation and gargling for the common cold. Sci Rep. 2019 Jan 31;9(1):1015. doi: 10.1038/s41598-018-37703-3. PMID 30705369
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen L, Liu HG, Liu W, Liu J, Liu K, Shang J, Deng Y, Wei S. [Analysis of clinical features of 29 patients with 2019 novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Feb 6;43(0):E005. doi: 10.3760/cma.j.issn.1001-0939.2020.0005. Online ahead of print. Chinese. PMID 32026671
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Sharma R, Hebbal M, Ankola AV, Murugaboopathy V, Shetty SJ. Effect of two herbal mouthwashes on gingival health of school children. J Tradit Complement Med. 2014 Oct;4(4):272-8. doi: 10.4103/2225-4110.131373. PMID 25379471
- [Background] Chatterjee A, Saluja M, Singh N, Kandwal A. To evaluate the antigingivitis and antipalque effect of an Azadirachta indica (neem) mouthrinse on plaque induced gingivitis: A double-blind, randomized, controlled trial. J Indian Soc Periodontol. 2011 Oct;15(4):398-401. doi: 10.4103/0972-124X.92578. PMID 22368367
- [Background] Chava VR, Manjunath SM, Rajanikanth AV, Sridevi N. The efficacy of neem extract on four microorganisms responsible for causing dental caries viz Streptococcus mutans, Streptococcus salivarius, Streptococcus mitis and Streptococcus sanguis: an in vitro study. J Contemp Dent Pract. 2012 Nov 1;13(6):769-72. doi: 10.5005/jp-journals-10024-1227. PMID 23404001
- [Background] Alzohairy MA. Therapeutics Role of Azadirachta indica (Neem) and Their Active Constituents in Diseases Prevention and Treatment. Evid Based Complement Alternat Med. 2016;2016:7382506. doi: 10.1155/2016/7382506. Epub 2016 Mar 1. PMID 27034694
- [Background] Badam L, Joshi SP, Bedekar SS. 'In vitro' antiviral activity of neem (Azadirachta indica. A. Juss) leaf extract against group B coxsackieviruses. J Commun Dis. 1999 Jun;31(2):79-90. PMID 10810594
- [Background] Arora R, Chawla R, Marwah R, Arora P, Sharma RK, Kaushik V, Goel R, Kaur A, Silambarasan M, Tripathi RP, Bhardwaj JR. Potential of Complementary and Alternative Medicine in Preventive Management of Novel H1N1 Flu (Swine Flu) Pandemic: Thwarting Potential Disasters in the Bud. Evid Based Complement Alternat Med. 2011;2011:586506. doi: 10.1155/2011/586506. Epub 2010 Oct 13. PMID 20976081
- [Background] Siddiqui BS, Ali SK, Ali ST, Naqvi SN, Tariq RM. Variation of major limonoids in Azadirachta indica fruits at different ripening stages and toxicity against Aedes aegypti. Nat Prod Commun. 2009 Apr;4(4):473-6. PMID 19475987
- [Derived] Burton MJ, Clarkson JE, Goulao B, Glenny AM, McBain AJ, Schilder AG, Webster KE, Worthington HV. Antimicrobial mouthwashes (gargling) and nasal sprays administered to patients with suspected or confirmed COVID-19 infection to improve patient outcomes and to protect healthcare workers treating them. Cochrane Database Syst Rev. 2020 Sep 16;9(9):CD013627. doi: 10.1002/14651858.CD013627.pub2. PMID 32936948
- [Derived] Khan FR, Kazmi SMR, Iqbal NT, Iqbal J, Ali ST, Abbas SA. A quadruple blind, randomised controlled trial of gargling agents in reducing intraoral viral load among hospitalised COVID-19 patients: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Sep 14;21(1):785. doi: 10.1186/s13063-020-04634-2. PMID 32928313
- See also: Burden of disease in COVID-19 pandemic — https://www.worldometers.info/coronavirus/
- See also: Recommendation on elective and cosmetic dental procedures by ADA — https://www.ada.org/en/publications/ada-news/2020-archive/march/ada-recommending-dentists-postpone-elective-procedures
- See also: Report on mortality of doctors and nurses combating corona virus pandemic — https://www.theguardian.com/world/2020/apr/16/doctors-nurses-porters-volunteers-the-uk-health-workers-who-have-died-from-covid-19